CLINICAL TRIAL: NCT02520635
Title: A Clinical Study of Supra-early Post-Surgery Chemotherapy Plus Standard TEMODAL® Regimen Versus Standard TEMODAL® Regimen in the Treatment on Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Supra-early Post-Surgery Chemotherapy in the Treatment on GBM Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Song Lin, Director of neurosurgical supratentorial tumor ward, Beijing Tiantan Hospital
Other Study IDs: B0008
Record Dates: First submitted 2015-06-26; First posted 2015-08-13 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Glioblastoma
Keywords: prognosis; supra-early chemotherapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TEMODAL® standard therapy regimen: 4 weeks after surgery, patients are administered with radiotherapy that consisted of fractionated focal irradiation at a dose of 2 Gy per fraction given once daily 5 dyas a week over a period of 6 weeks. Concomitant TEMODAL® are administered orally at a daily dose of 75mg/m2 from the first day of radiotherapy until the last day of radiotherapy, but for no longer than 49 days. After a 4-week break, patients were then to receive up to 6 cycles of adjuvant TEMODAL® chemotherapy according to the standard 5-day schedule every 28 days.The dose is 150mg/m2 once daily for cycle 1 and is increase to 200mg/m2 at the beginning of cycle 2, so long as there were no hematologic toxic effects.
  Interventions: Drug: standard TEMODAL® chemotherapy; Radiation: Radiotherapy 60Gy
- post-surgery supra-early TEMODAL® chemotherapy: Within 24 hours after surgery, Supra-early TEMODAL® Chemotherapy is administered orally at 75mg/m2/day for 28 days for patients pathologically confirmed as GBM. 4 weeks after surgery, patients are administered with radiotherapy that consisted of fractionated focal irradiation at a dose of 2 Gy per fraction given once daily 5 dyas a week over a period of 6 weeks. Concomitant TEMODAL® are administered orally at a daily dose of 75mg/m2 from the first day of radiotherapy until the last day of radiotherapy, but for no longer than 49 days. After a 4-week break, patients were then to receive up to 6 cycles of adjuvant TEMODAL® chemotherapy according to the standard 5-day schedule every 28 days.The dose is 150mg/m2 once daily for cycle 1 and is increase to 200mg/m2 at the beginning of cycle 2, so long as there were no hematologic toxic effects.
  Interventions: Drug: supra-early TEMODAL® chemotherapy; Radiation: Radiotherapy 60Gy

INTERVENTIONS:
Drug: supra-early TEMODAL® chemotherapy
  Groups: post-surgery supra-early TEMODAL® chemotherapy
Drug: standard TEMODAL® chemotherapy
  Groups: TEMODAL® standard therapy regimen
Radiation: Radiotherapy 60Gy

SUMMARY:
The primary purpose of the study is to evaluate the efficacy and safety of supra-early post-surgery chemotherapy versus standard TEMODAL® regimen in treatment of patients with newly diagnosed glioblastoma multiforme. The secondary purpose is to assess the efficacy of supra-early post-surgery chemotherapy in release brain edema.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common primary malignant brain tumor. Despite great efforts have been devoted to promoting the treatment effect, GBM remains one of the most lethal tumors concurrent with poor prognosis and inevitable recurrence. The standard treatment protocol for GBM includes surgical resection, radiotherapy and temozolomide (TMZ) based chemotherapy. TMZ, an alkylating agent, has been proved to be efficient to control tumor growth after surgery and gradually has been recognized in routine clinical course for GBM. In a pivotal clinical trial published in 2005, GBM patients received concomitant TMZ and radiotherapy followed by 6 periods of adjuvant TMZ chemotherapy had a median survival of 14.6 months and 5-year survival rate of 9.8%, which has been regarded as a landscape in treatment history of GBM. To date, this regimen remains the standard protocol for newly diagnosed GBM patients. However, the optimal timing of initiation of TMZ or radiotherapy remains unclear. Our previous study showed 75mg per square meter of body surface per day (mg/m2/d) of TMZ chemotherapy alone was effective to control post-operative edema caused by tumor cell infiltration in primary GBM patients. The result suggested anti-cancer agents such as TMZ may be a useful regimen to control tumor cell regrowth after operation. Therefore, we conducted this prospective clinical trial to testify the hypothesis that supra-early initiation of TMZ chemotherapy in newly diagnosed GBM patients is effective to control tumor growth after tumor resection and therefore improve patients'clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with prior histological confirmation of newly diagnosed primary glioblastoma multiforme in supratentorial cerebral hemisphere.
2. Gross total resection or partial resection (imaging) >70%.
3. Chemo-radiotherapy to be expected from Week 5 (Day 29) after surgery.
4. Age >=18 and <=70 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
6. Life expectancy >=9 months.
7. Laboratory test values must satisfy the following criteria:

   1. absolute neutrophil count >=1.5 x 10^9/L;
   2. platelet count >=100 x 10^9/L;
   3. hemoglobin >=80 g/L;
   4. blood urea nitrogen and creatinine < 1.5 x upper limit of normal value (ULN);
   5. total bilirubin and direct bilirubin < 1.5 x ULN;
   6. alanine aminotransferase and aspartate aminotransferase < 3 x ULN;
   7. alkaline phosphatase < 2 x ULN.
8. Patients must be willing to provide written informed consent.
9. Patients of child-bearing potential (including female subjects and the female partners of male subjects) must use an effective method of contraception.

Exclusion Criteria:

1. Patients without prior histological confirmation of primary glioblastoma multiforme.
2. Patient with previous or current malignancies at other sites.
3. Patient who received chemotherapy, radiotherapy for study indication, or other medications for antitumor indication prior to surgery.
4. Patient with recurrent or multiple malignant glioma (including gliomatosis cerebri).
5. Patient with metastatic lesions at the subtentorial or outside of calvaria.
6. Patient who received chemotherapy or radiotherapy sensitizers for head or neck tumor.
7. Patient who received radiotherapy at head or neck which leads to radiotherapy domain overlapping.
8. Frequent vomiting or medical condition that could interfere with oral medication intake (eg, partial bowel obstruction).
9. Known human immunodeficiency virus (HIV)-positive or acquired immune deficiency syndrome (AIDS)-related illness.
10. Woman who is pregnant or breastfeeding.
11. Patient with a history of hypersensitivity to temozolomide or other analogic alkylating agents.
12. Patient with severe myelosuppression
13. Patient with any other conditions under which investigators think the subject is not suitable for enrolment, such like having known that the subject may not have good compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prior histological confirmation of newly diagnosed primary glioblastoma multiforme in supratentorial cerebral hemisphere.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | Up to 2 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 2 years
Objective Response Rate | Up to 2 years
Treatment-related adverse event | Up to 2 years
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Song Lin, MD, Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China